CLINICAL TRIAL: NCT03340558
Title: A Pilot Study Investigating the Effect of Atezolizumab Monotherapy and Atezolizumab Plus Cobimetinib on the Tumoral Immunoprofile in Liver Metastases From Colorectal Cancer
Brief Title: Atezolizumab Monotherapy vs Atezolizumab Plus Cobimetinib in Liver Metastases From Colorectal Cancer
Acronym: ATELIER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Negative results in a similar study
Sponsor: Niharika Mettu (Other)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor-Investigator, Niharika Mettu, Medical Instructor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00085578
Record Dates: First submitted 2017-11-09; First posted 2017-11-13 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — atezolizumab; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy Cohort (Experimental): The first 10 subjects will receive Atezolizumab 840 mg IV on Day 1 and Day 15 of each 28-day cycle. Subjects will be treated for 2 cycles before undergoing metastatectomy within 42 days of completion of Cycle 2. No study treatment is administered while subjects are healing after surgery.
  Interventions: Biological: Atezolizumab
- Combination Cohort (Experimental): The next 15 subjects will receive Atezolizumab 840 mg IV on Day 1 and Day 15 and Cobimetinib 60 mg PO on Days 1-21 of each 28-day cycle. Cobimetinib must be held for the 7 days prior to metastatectomy. Subjects will be treated for 2 cycles before undergoing metastatectomy within 42 days of completion of Cycle 2.
  Interventions: Biological: Atezolizumab; Drug: Cobimetinib

INTERVENTIONS:
Biological: Atezolizumab — Atezolizumab is a fully humanized, engineered monoclonal antibody of IgG1 isotype against the protein programmed cell death-ligand 1.
Drug: Cobimetinib — MEK inhibitor
  Arms: Combination Cohort

SUMMARY:
This study is for patients with metastatic colorectal cancer who are candidates for resection of metastases. This study will be conducted sequentially with 2 cohorts: 1.) Monotherapy Cohort and 2.) Combination Cohort

Pre-metastatectomy

* Monotherapy Cohort: The first 10 subjects will receive Atezolizumab 840 mg IV on Day 1 and Day 15 of each 28-day cycle.
* Combination Cohort: The next 15 subjects will receive Atezolizumab 840 mg IV on Day 1 and Day 15 and Cobimetinib 60 mg PO on Days 1-21 of each 28-day cycle. Note: Cobimetinib must be held for the 7 days prior to metastatectomy.

All subjects will be treated for 2 cycles (8 weeks) prior to metastatectomy

Metastatectomy

Subjects will undergo liver metastatectomy within 42 days of completion of Cycle 2 of pre-metastatectomy treatment. No study treatment is administered while the patient is healing after surgery.

Post-metastatectomy

Once the patient has healed from the surgery, adjuvant treatment may be administered at the discretion of the treating physician. Restaging following standards of care for this setting.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed and radiographically measurable per RECIST v1.1 colorectal cancer with liver metastasis. Patients may have other sites of metastatic disease.µlµ
2. Liver lesion safely amenable to core needle biopsy.
3. Willing to undergo core needle biopsy of liver metastatic site.
4. Microsatellite stable disease as determined by IHC and/or PCR.
5. Plan for next therapeutic intervention to be surgical resection of metastatic disease.
6. Age ≥18 years with ability to understand and willingness to provide informed consent.
7. ECOG performance status of 0 or 1.
8. Life expectancy of >3 months.
9. For Combination Therapy cohort only: Able to swallow pills.
10. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to start of study drug and must be willing to use two methods of contraception, one of them being a barrier method during the study and for 3 months (or 6 months for subjects on Combination Therapy cohort) after last study drug administration.
11. Adequate organ and marrow function as defined below:

    1. Absolute neutrophil count (ANC) ≥1500 µl
    2. WBC counts > 2500/µl
    3. Lymphocyte count ≥ 300/µl
    4. Platelets ≥ 100,000/µl
    5. Hemoglobin (Hgb) ≥ 9 g/dL
    6. Total bilirubin ≤ 1.5 x upper limit of normal (ULN); ≤ 3 x ULN for patients with known Gilbert disease
    7. AST/ALT ≤ 3 x ULN without liver metastasis; ≤ 5 x ULN for patients with liver metastasis
    8. Alkaline phosphatase ≤ 2.5 x ULN; ≤ 5 x ULN for patients with liver metastasis
    9. Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 ml/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation
    10. INR and aPTT ≤ 1.5 x ULN. Note that this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose.

Exclusion Criteria:

1. Prior therapy with anti-PD-1 or anti-PD-L1 therapeutic antibody or pathway targeting agents.

   a. Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met: i. Minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose.

   ii. No history of severe immune-related adverse effects from anti-CTLA-4 (NCI CTCAE Grade 3 and 4)
2. For Combination Therapy cohort only: Prior therapy with MEK inhibitors.
3. Anticancer therapy, including but not limited to chemotherapy, hormonal therapy, or radiotherapy, within 4 weeks prior to start of study treatment; however, the following are allowed:

   1. Hormone-replacement therapy or oral contraceptives
   2. Herbal therapy > 1 week prior to start of study treatment (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to start of study treatment)
   3. Palliative radiotherapy for bone metastases > 2 weeks prior to start of study treatment
4. Expected to require any other form of systemic or localized anticancer therapy while on study.
5. Adverse events from prior anticancer therapy that have not resolved to Grade ≤ 1 except for alopecia.
6. Investigational agent within 4 weeks prior to start of study treatment (or within five half-lives of the investigational product, whichever is longer).
7. Major surgical procedure within 28 days prior to start of study treatment or anticipation of need for a major surgical procedure during the course of the study. This does not refer to the planned liver metastatectomy that is part of the study.
8. Malignancies other than the disease under study within 5 years prior to start of study treatment, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g. chronic lymphocytic leukemia Rai stage 0, prostate cancer with Gleason score < 6, and prostate-specific [PSA] ≤ 10 mg/mL, etc).
9. Diagnosis of acute leukemias, accelerated/blast-phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma.
10. Prior allogenic bone marrow transplantation or prior solid organ transplantation.
11. Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases.

    a. Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met: i. Evaluable or measurable disease outside the CNS ii. No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm) iii. No history of intracranial hemorrhage or spinal cord hemorrhage iv. No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted.

    v. No neurosurgical resection or brain biopsy within 28 days prior to start of study treatment b. Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following: i. Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study ii. No stereotactic radiation or whole-brain radiation within 28 days prior to start of study treatment iii. Screening CNS radiographic study ≥ 4 weeks from completion of radiotherapy and ≥ 2 weeks from discontinuation of corticosteroids
12. Serious, non-healing wound, ulcer, or bone fracture.
13. Pregnancy, lactation, or breastfeeding
14. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins or Chinese hamster ovary cell products.
15. History of malabsorption or other condition that would interfere with absorption of cobimetinib.
16. Bisphosphonate therapy for symptomatic hypercalcemia. Use of bisphosphonate therapy for other reasons (e.g., bone metastasis for osteoporosis) is allowed.
17. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease.
18. History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis.

    1. Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone, controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible.
    2. Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    i. Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations ii. Rash must cover less than 10% of the body surface area (BSA) iii. Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%) iv. No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation (PUVA), methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
19. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. (History of radiation pneumonitis in the radiation field (fibrosis) is permitted)
20. Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]-α or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to start of study treatment.
21. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to start of study treatment.

    1. Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
    2. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
22. History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection

    1. Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
    2. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
23. Active tuberculosis
24. Severe infections within 4 weeks prior to start of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
25. Signs or symptoms of infection within 2 weeks prior to start of study treatment
26. Received oral or IV antibiotics within 2 weeks prior to start of study treatment

    a. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
27. Administration of a live, attenuated vaccine within 4 weeks before start of study treatment or anticipation that such a live, attenuated vaccine will be required during the study

    a. Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to start of study treatment or at any time during the study.
28. History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, retinal vein occlusion (RVO), or neovascular macular degeneration. Patients should be excluded if they have the following risk factors for RVO:

    1. History of serous retinopathy
    2. History of retinal vein occlusion (RVO)
    3. Evidence of ongoing serous retinopathy or RVO at baseline
29. History of clinically significant cardiac dysfunction, including the following:

    1. Current unstable angina
    2. Current symptomatic congestive heart failure of NYHA class 2 or higher
    3. Uncontrolled hypertension ≥ Grade 2 (patients with a history of hypertension controlled with anti-hypertensives to ≤ Grade 1 are eligible).
    4. Left ventricular ejection fraction (LVEF) below institutional LLN or below 50%, whichever is lower
    5. Uncontrolled arrhythmias
    6. Myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack within the previous 6 months
30. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results of render the patient at high risk from treatment complications.
31. Inability to comply with study and follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in CD4 T cell immune infiltrates | Subject tissue will be assessed pre-treatment (baseline) and post-treatment within 42 days after completion of Cycle 2 using metastatectomy tissue.
  The change in CD4 T cell tumor infiltrates will be measured as the absolute number of infiltrates per number of high-powered fields. The paired t-test will be used to compare changes in CD4 T cells in pre- and post-treatment.
Change in CD8 T cell immune infiltrates | Subject tissue will be assessed pre-treatment (baseline) and post-treatment within 42 days after completion of Cycle 2 using metastatectomy tissue.
  The change in CD8 T cell tumor infiltrates will be measured as the absolute number of infiltrates per number of high-powered fields. The paired t-test will be used to compare changes in CD8 T cells in pre- and post-treatment.

SECONDARY OUTCOMES:
Disease-free survival | Disease-free survival will be measured from study entry up to 5 years.
  The length of time after primary treatment that the subject survives without any signs or symptoms of that cancer.
Overall Survival | Overall survival will be measured from study entry up to 5 years
  The length of time from start of treatment that the subject is alive

CONTACTS AND LOCATIONS:
Overall Officials: Niharika Mettu, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States